CLINICAL TRIAL: NCT05724381
Title: Auramine Phenol Staining Technique for Revealing Different Coccidian Parasites
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khoulood Zakaria Hashem, Assistant lecturer of medical parasitology at the Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-23-01-25
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Chronic Diarrhea
Keywords: coccidian parasites; auramine phenol staining; fluorescence microscopy; modified Ziehl Nelseen; Cryptosporidium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: auramine phenol staining — The samples will be divided into 2 parts. The 1st part will be subjected to a direct wet saline smear, iodine smear, and concentration techniques. The 2nd part will be used to perform thin smears of the fecal concentrates and air-dried on 2 different slides. The first slide will be stained with Kinyoun's acid-fast stain and examined with the conventional light microscope and the second will be stained with auramine-phenol stain and examined with the fluorescent microscope.

SUMMARY:
The increased number of documented human coccidian infections, including Cryptosporidium parvum, Cyclospora cayetanensis, Isospora belli, and Sarcocystis spp., that are often indistinguishable from other forms of community-acquired diarrhea, together with the possibility of treating some of them, suggests a need for proper diagnostic techniques to recover and identify these organisms

DETAILED DESCRIPTION:
The increased number of documented human coccidian infections, including Cryptosporidium parvum, Cyclospora cayetanensis, Isospora belli, and Sarcocystis spp., that are often indistinguishable from other forms of community-acquired diarrhea, together with the possibility of treating some of them, suggests a need for proper diagnostic techniques to recover and identify these organisms.

Earlier, Cryptosporidium and Cystoisospora were assumed to be the causative agents of acute diarrhea in animals but recently have emerged as one of the leading causes of prolonged lifethreatening diarrhea in immunocompromised patients particularly in those with immune dysfunction like AIDS who may show severe intestinal injury, prolonged diarrhea, extreme weight loss, and generalized wasting. In contrast, healthy individuals commonly present with mild to moderate self-limiting diarrhea during the infective stage, besides asymptomatic infection can also occur.

Detection of coccidian parasites is mostly through microscopic observation using Kinyon's acid-fast stain. Although Sheather sugar flotation may result in increased concentration of the cysts, this method is cumbersome and does not lend itself to convenient incorporation within the routine concentration and staining procedures favored in most clinical laboratories. Any acid-fast stain will be taken up by cyst walls, but the time required to prepare and examine acid-fast stains on all stool samples received for routine parasitology would not be cost-effective unless the prevalence of coccidian parasites was shown to warrant such effort.

ELIGIBILITY:
Inclusion Criteria:

* patients complaining of chronic diarrhea .

Exclusion Criteria:

* patients taking antibiotics within the previous four weeks, and anti-parasitic drugs within the previous two weeks.

Ages: 6 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients from outpatient clinics in different hospitals in Sohag governorate complaining of diarrhea of any age and sex groups from different locations (cities and villages)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of coccidian parasites | 1 month
  number of patients positive for coccidian parasites

SECONDARY OUTCOMES:
auramine phenol staining | 1 month
  accuracy of auramine phenol staining in the detection of coccidian parasites in comparison to light microscopy

IPD SHARING:
Plan to Share IPD: Undecided